CLINICAL TRIAL: NCT02976090
Title: Phenotyping of Small Bowel Adenocarcinoma
Acronym: BIONADEGE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); Centre Hospitalier Universitaire de Besancon (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Other Study IDs: NI14026
Record Dates: First submitted 2016-10-25; First posted 2016-11-29 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2018-11

CONDITIONS: Small Bowel Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumour block
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the fact that small intestine makes up 75% of the length of the digestive tract and 90% of its mucosal surface area, small bowel adenocarcinoma (SBA) is rare. SBA is not equally dispatched along the small bowel, a predisposing disease is frequently associated. All these data suggest particular carcinogenesis pathway. SBA carries poor prognosis at all stages and no standard treatment have proved efficacy. So far, no data are available for targeted therapy. From the literature and a previous study of our group some biologic data showed that SBA carcinogenesis is closer to colorectal than gastric carcinogenesis. Nevertheless, some differences arise (ie: low Adenomatous Polyposis Coli mutation rate or frequent DNA mismatch repair deficiency). Even if some trends are founded the prognostic value of molecular alteration and phenotype variation according to small bowel segment, or predisposing disease could not been demonstrate due to small sample size.

BIONADEGE study is a planned biologic ancillary study of the NADEGE cohort that enrolled 366 patients with SBA from 2009 to 2012 in France. The tumour blocks and clinical data of 187 patients have been collected. The main objective is to assess the prognostic value for recurrence free survival (RFS) in non-metastatic patients and overall survival (OS) in metastatic patients of molecular alteration in a set of 46 genes and abnormal protein expression potentially implicated in carcinogenesis. The mains secondary objectives are: 1) to identify potential mutation targetable in small intestine tumours and protein expression, 2) to state the frequency of molecular alteration according to the tumour location, stage or predisposing disease and established clinico-biologic correlation. Tissue microarrays will be performed and several potential prognostic markers will be assessed. Sequencing on tumour DNA will investigate the presence of 740 hot spot somatic mutations in 46 genes involved.The abnormal protein expression or the genetic alterations with an expected frequency superior to 10% will be assessed as potential prognostic factor to RFS and OS.

These evaluations on a large cohort could allow comparison between pathways and will offer better knowledge of tumour molecular phenotype and prognosis will give rational for targeted therapy trials The predisposing diseases for SBA involved several different carcinogenesis pathways. Finally, a molecular classification of SBA will be attempt.

DETAILED DESCRIPTION:
The NADEGE cohort involves 75 centres and had enrolled 365 patients. Among them 232 patients had a resection of the primary tumour in 58 centres. This will is be the largest series in the world of SBA for biological study. The patients enrolled in the NADEGE cohort were aware of the biologic study and their authorisation to perform is already collected.

Baseline clinical data of patients enrolled in NADEGE cohort are already available and were presented in a poster discussion session at the European Society for Medical Oncology congress 2013. In all the cohort the primary location was duodenum in 51% of the patients, and a predisposing disease was reported in 18.8% of the patient mainly Crohn disease in 8% and Lynch syndrome in 6% of the patients. The follow-up is ongoing. The analyses of 3-years recurrence-free survival is planned in 2015 and the analysis of 5-years overall survival in 2017.

Today 187 tumour sample are collected and archived in the pathology department of Saint Antoine hospital (Paris). Among these 187 tumours the tumour stage are: stage 0: 4, stage I: 10, stage II: 34, stage III: 63, undetermined stage non-metastatic: 30 (thus 141 non-metastatic tumours) and stage IV: 48, and the primary are: duodenum: 128, jejunum: 31, ileon: 27, undetermined: 3. The chemotherapy performed was FOLFOX in 80% of the cases.

Work Package 1: Database (team 1) The clinical data of NADEGE cohort are collected with an e-crf. The initial descriptive data are already monitored by the GERCOR team. The results have been already presented. BIONADEGE is a planned ancillary study of the NADEGE cohort. The complementary queries for the purpose of BIONADEGE will be addressed by the team 1 to the NADEGE investigator. The follow-up data for progression (metastatic patients), recurrence (non-metastatic patient) and death (all patients) will be obtained every 6 months. Follow-up data will be collected until 2019 in order to obtain 5-years follow-up for all the patients.

Work Package 2: Anatomopathology (team 2) All the tumour samples are already bank in the pathology laboratory of Saint Antoine hospital. Slides from representative tumour area will be selected and send to Paris Descartes university to allow DNA extraction. Tissue microarrays (TMA) for immunohistochemistry validation studies will be performed. Several potential prognostic markers will be assessed as MismatchRepair (MMR) protein, P53, beta-catenin, c-myc protein. Other predictive markers for chemotherapy as hENT1, O6-methylguanine DNA methyltransferase (MGMT) and for targeted therapy as Proto-oncogene tyrosine-protein kinase (ROS1), hepatocyte growth factor receptor c-Met (HGFR), Alk, Human Epidermal Growth Factor Receptor-2 (HER-2) and Programmed cell death 1 (PD-1) will also be assessed. The cases overexpressing HER-2 and HGFR protein by immunohistochemistry will be tested by Fluorescent In Situ Hybridisation (FISH).

Work Package 3: Biochemistry (team 3) DNA will be extracted from tumour block in the university unit S1147 according to the following protocol. Using a 1.0-mm punch, paraffin embedded tissues from all cases will be sampled from representative areas that will contain more than 50% of tumour cells. DNA will be thereafter extracted from each sample following the manufacturer's recommendation. The team3 will use a competitive allele specific taqman probe designed on Kras wild type allele (Hs.00000174-rf - Life Technologies) on serial dilution of each DNA sample in order to quantify amplifiable DNA. Only samples with more than 10 ng of amplifiable DNA will be retained for the sequencing. DNA from each sample will be amplified. The presence of more than 740 hot spot somatic mutations in the 46 genes will be investigate. Data analysis, including alignment to the hg19 human reference genome and variant calling, will be done using the Software of Life Technologies. Alignments will be visually verified and annotated with the software of Integrative Biosoftware. A sequence variation will be considered as a potential mutation if (i) the coverage is superior to 200×, (ii) the allelic frequency is superior to 10%, (iii) the strand bias is from 0.2 to 0.8, (iv) the variation is not reported in the 1000 genomes database, (v) the variation is a missense or a non-sense variation. All these selected variations will be controlled using the Sanger sequencing technics using amplified fragments of less than 150 bp centred on the potential mutation.

ELIGIBILITY:
Inclusion Criteria:

* patients included in NADEGE cohort
* patients with available and exploitable biological samples from NADEGE cohort

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients included in NADEGE cohort
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
RFS in non-metastatic patients according to 46 genes and abnormal protein expression potentially implicated in carcinogenesis. | 3 years

SECONDARY OUTCOMES:
OS in metastatic patients according to 46 genes and abnormal protein expression potentially implicated in carcinogenesis | 3 years
Rate of MMR status | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sabine HELFEN, Study Chair — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aparicio T, Svrcek M, Henriques J, Afchain P, Lievre A, Tougeron D, Gagniere J, Terrebonne E, Piessen G, Legoux JL, Lecaille C, Pocard M, Gornet JM, Zaanan A, Lavau-Denes S, Lecomte T, Deutsch D, Vernerey D, Puig PL. Panel gene profiling of small bowel adenocarcinoma: Results from the NADEGE prospective cohort. Int J Cancer. 2021 Apr 1;148(7):1731-1742. doi: 10.1002/ijc.33392. Epub 2021 Jan 4. PMID 33186471